CLINICAL TRIAL: NCT06156826
Title: Baseline Nutritional Status During Pregnancy
Brief Title: Prenatal Nutrient Status Study
Status: Completed | Type: Observational
Sponsor: Needed PBC (Industry)
Responsible Party: Sponsor
Other Study IDs: ND.001
Record Dates: First submitted 2023-11-15; First posted 2023-12-05 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy Related; Nutrient Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research is to gather data on nutritional status from approximately 250 pregnant women who are currently taking a prenatal vitamin in order to better understand if the prenatal vitamins that most people use are providing enough nourishment during pregnancy.

Participants will be asked to:

* complete an online survey
* schedule a blood draw for the Study Multivitamin Blood Test
* complete the blood draw visit
* complete a final survey at study end

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speaks, reads, and understands English
* Lives in the United States
* Lives within a ZIP code from the metropolitan areas where mobile phlebotomists will be available for blood draws
* Assigned female sex at birth
* Currently within weeks 24-34 of pregnancy
* Currently taking a daily prenatal vitamin

Exclusion Criteria:

* Birth sex other than female
* Currently taking a prenatal vitamin without Folic Acid other than Needed Prenatal Multivitamin

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who are currently pregnant who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-08-24 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Percentage of sample deficient in each nutrient in pregnant women | Baseline
  Stratified by the type of prenatal vitamin they are taking at baseline (standard or Needed Prenatal Multivitamin).

CONTACTS AND LOCATIONS:
Overall Officials: Ari Calhoun, ND, Principal Investigator — Wholesome Brain Medicine
Locations (1):
- Needed PBC, Los Angeles, California, United States